CLINICAL TRIAL: NCT06343480
Title: Sublingual Misoprostol Versus Oxytocin Titration for Induction of Labour in Parturients With Spontaneous Rupture of Fetal Membranes at Term: A Randomised Controlled Tial.
Brief Title: Misoprostol Versus Oxytocin for Induction of Labour in Parturients With Spontaneous Rupture of Fetal Membranes at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Nwali Matthew Igwe, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMVOT2024CT
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Labor Onset and Length Abnormalities
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first arm - Oxytocin titration (Active Comparator): Received vitamin c 100mg as placebo and had Oxytocin titration in 500ml of ringers lactate for labour induction
  Interventions: Drug: Labour Induction
- second arm - Misoprostol give sublingual (Active Comparator): received 25mcg of Misoprostol and titration of plane 500ml of ringers lactate as placebo
  Interventions: Drug: Labour Induction

INTERVENTIONS:
Drug: Labour Induction — the use of misoprostol sublingual for labour induction compared with oxytocin titration in parturients with prelabour membrane rupture at term.
  Other Names: oxytocin titration

SUMMARY:
Intravenous oxytocin titration has a prime position as a choice agent for induction of labour following term PROM as it has been shown to be efficacious for such purpose. Recent evidence however has shown that misoprostol is associated with better outcomes and merits evaluation in our environment. This study compared the efficacy of misoprostol and oxytocin for induction of labour in parturients with term Prelabour Ruptuture of Membranes.

DETAILED DESCRIPTION:
Induction of labour for term premature rupture of fetal membranes (PROM) is associated with greater maternal satisfaction and lower risk of maternal infection compared with expectant management. The ideal method of induction of labour for term PROM is a subject of controversy. Intravenous oxytocin titration has a prime position as a choice agent for induction of labour following term PROM as it has been shown to be efficacious for such purpose. Recent evidence however has shown that misoprostol is associated with better outcomes and merits evaluation in our environment.

This study compared the efficacy of misoprostol and oxytocin for induction of labour in parturients with term PROM. This was a double blind randomized controlled trial on the efficacy of sublingual misoprostol versus oxytocin titration in women with term PROM at the Alex Ekwueme Federal University Teaching Hospital Abakaliki (AEFUTHA) and Mile 4 Hospital Abakaliki. 240 Participants were divided into two groups of 120 participants each. Group A received 25 mcg of sublingual misoprostol and titration of 500 ml of Ringer's lactate solution as placebo with 5ml of sterile water injected into it while group B underwent immediate induction of labour with titration of 5 units of oxytocin in a 500 ml of Ringer's lactate solution and received one tablet of 100mg Vitamin C as placebo. The primary outcome measure was the mean induction delivery interval. The secondary outcome measures were Caesarean section rate, the incidence of uterine hyper-stimulation, tachysystole or hypertonus, APGAR scores at the first and fifth minute and NICU admission. Data analysis was done using statistical Package for Social Science (IBM SPSS) software (version 20, Chicago IL, USA). Continuous variables were presented as mean and standard deviation (Mean ± SD), while categorical variables were presented as numbers and percentages. Categorical variables were analyzed using Chi-square while means were compared using T-test. A difference with a P value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* singleton pregnancy at term
* prelabour rupture of membranes
* not having contraction
* Bishop scoe 5 or less

Exclusion Criteria:

* prelabour rupture of membranes at less than term
* declined consent
* contraindication for vaginal delivery
* multiple gestation
* medical conditions co-existing with pregnancy
* grand multiparous parturients
* previous caesarean section scar
* already having contractions
* has intrauterine foetal death
* bishop sore >5

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Mean induction delivery interval | During the delivery
  the time take from start of induction to the time of delivery of the fetus.

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State
  - Federal Teaching Hospital, Abakaliki, Abakaliki, Ebonyi State